CLINICAL TRIAL: NCT03105700
Title: Safety and Feasibility of Accelerated Low-Frequency Transcranial Magnetic Stimulation for Medication-Resistant Depression in Patients With Epilepsy
Brief Title: Low Frequency TMS for Depression in Epilepsy
Acronym: LFTMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: The Diamond Foundation Inc. (Other)
Responsible Party: Principal Investigator, Krzysztof Bujarski, Staff Physician, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D16150
Record Dates: First submitted 2017-03-06; First posted 2017-04-10 (Actual); Results first posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Epilepsy; Depressions, Refractory
Keywords: epilepsy; depression; refractory; TMS
MeSH Terms: conditions — Epilepsy; Depressive Disorder, Treatment-Resistant; Depression | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Low Frequency TMS Intervention (Experimental): Patients will receive low-frequency TMS on an accelerated schedule over three consecutive days.
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — Repetitive transcranial magnetic stimulation (TMS) is a focal, nonpharmacological, noninvasive method for stimulating the brain and modulating neural network activity. To administer TMS, an electromagnetic coil is placed on the scalp, and uses electrical current to create magnetic fields that depolarize or hyperpolarize neurons in the brain.
  Other Names: Mag-Venture Mag-pro; TMS

SUMMARY:
The purpose of this study is to determine if low-frequency transcranial magnetic stimulation (TMS) is safe and feasible for treating depressive symptoms in patients with epilepsy. Patients will receive an accelerated protocol of TMS consisting of three consecutive days of treatment. Patients will have in-person follow up visits after one month and again after six months.

DETAILED DESCRIPTION:
This is a pilot study designed primarily to assess whether patients with epilepsy can safely tolerate low-frequency transcranial magnetic stimulation in an accelerated protocol to treat depression. The investigators aim to treat 12 patients with epilepsy and comorbid depression to receive a total of 15 hours of transcranial magnetic stimulation over 3 days at Dartmouth-Hitchcock Medical Center (DHMC). The investigators will assess safety of this protocol with regards to seizure frequency and other side effects of TMS treatment and the feasibility of using an accelerated protocol in this patient population. In addition to these primary aims, our secondary goal is to determine if dense array EEG can provide a useful biomarker for depression and its treatment in focal epilepsy. A structural and functional MRI will be obtained before treatment and a dense array EEG before and after TMS treatment to assess for changes in specific dense array EEG based biomarkers.

In addition to recruiting patients, the study staff will likewise request that family members or friends of the patient accompany the patient monitor him/her for increased seizure frequency. The recruited family member will bring the patient to the treatment and stay with the patient overnight at a local hotel and monitor for possible seizures or other adverse events of treatment. Family members will be instructed in seizure safety and be given emergency phone numbers to call if the patient is experiencing adverse effects of TMS.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Able and willing to provide informed consent.
* Diagnosis of epilepsy confirmed by the study neurologist (KB).
* English-speaking
* Not pregnant
* Able to safely undergo MRI (as assessed by MRI safety form).
* Have a family member or friend (proxy) who will be able to bring the patient to the hospital and serve as a safety monitor during stay in study hotel for two consecutive nights.
* Patients on stable doses of current antiepileptic and antidepressant medications for 1 month.

Exclusion Criteria:

* Significant cognitive impairment measured by the Montreal Cognitive Assessment (MOCA) <23.
* History of other major psychiatric disorders (e.g., schizophrenia, bipolar disorder, substance use disorder (except caffeine and nicotine) or presence of unstable medical comorbidities.
* Actively/imminently suicidal (QIDS item 12 score > 2 or Mini-International Neuropsychiatric Interview (MINI) Suicidality module score > 16)
* Greater than 10 seizures per week during 1 month prior.
* History of stroke, moderate-severe traumatic brain injury or other major neurological disorder.
* Any magnetic or implanted device that will interfere with ability to safely receive MRI and/or TMS treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Krzysztof A. Bujarski, MD, Principal Investigator — Associate Professor of Neurology
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be de-identified and then available upon request from PI.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low Frequency TMS Intervention
Started | 15
Completed | 8
Not Completed | 7
Not completed — screen fail | 3
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Population: Patients that were enrolled.
Arm/Group | Low Frequency TMS Intervention
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants] — Population: 3 prospective participants were screen fails
  Participants
    number analyzed (Participants) | 12
    <=18 years | 0
    Between 18 and 65 years | 12
    >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 3 prospective participants were screen fails
  Participants
    number analyzed (Participants) | 12
    Female | 8
    Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 3 prospective participants were screen fails
  Participants
    number analyzed (Participants) | 12
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 12
    More than one race | 0
    Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants] — Population: 3 prospective participants were screen fails
  participants
    United States: number analyzed (Participants) | 12
    United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Seizure Frequency Expressed as the Average Number of Seizures Experienced by All Participants and Recorded at Specified Time Points Throughout the Study.
Description: The hypothesis is that TMS treatment will not produce serious adverse events defined as an increase in the average number of seizures across all participants. This data is collected from the time of enrollment, and then at baseline, 1-week post treatment, 1-month post-treatment, and 6-month post treatment. The seizures are reported directly by the participants during check-ins with the research staff at the study specified study timepoints.
Time Frame: Baseline, 1-week post-treatment, 1-month post-treatment, 6-month post-treatment follow-up
Population: Subjects 3 and14 were lost to 6-month follow-up for unknown reasons. Subjects 9 and 13 were lost to 6-month follow-up due to COVID 19.
Measure: Mean (Full Range); unit: average number of seizures
Arm/Group | Low Frequency TMS Intervention
Number analyzed (Participants) | 12
average number of seizures
  Baseline | 5.83 [0 to 40]
  1-week post-treatment | 0 [0 to 0]
  1-month post-treatment | 1.42 [0 to 12]
  6-month post-treatment: number analyzed (Participants) | 8
  6-month post-treatment | 1.0 [0 to 6]

2. Primary Outcome: Percentage of Participants Who Complete the TMS Treatment
Description: The percentage of participants who completed the TMS treatment as measured by the total number of participants (expressed as percentage) who completed 15-hour sessions of TMS over 3 days.
Time Frame: 15 one-hour sessions of TMS over 3 days
Population: Participants who started the TMS treatment and completed all sessions
Measure: Count of Participants; unit: Participants
Arm/Group | Low Frequency TMS Intervention
Number analyzed (Participants) | 12
Participants | 12

3. Primary Outcome: Number of Treatment-emergent Adverse Events as Measured by a Modified Systematic Assessment for Treatment Emergent Events (SAFTEE).
Description: The hypothesis is that TMS treatment will not be associated with a higher rate of adverse events as measured by a modified Systematic Assessment for Treatment Emergent Events (SAFTEE) given pre-TMS treatment and immediately post-TMS sessions. SAFTEE is a tool used to assess participants' adverse events and is presented to all participants before and right after each TMS session. The outcome is expressed as a total number of adverse events across all participants and all TMS treatment sessions.
Time Frame: Day 1, 2, and 3 of TMS treatment
Measure: Number; unit: adverse events
Arm/Group | Low Frequency TMS Intervention
Number analyzed (Participants) | 12
adverse events | 1

4. Primary Outcome: Measuring Biomarker for Depression Using Dense-array EEG
Description: Examine the utility of dense-array electroencephalogram (EEG) as a biological marker (biomarker) of depression and response to treatment with low-frequency transcranial magnetic stimulation (TMS) in patients with Epilepsy. The ratio of alpha power between the right and the left hemispheres is considered an EEG based biomarker for depression. It is obtained by dividing alpha power from the right brain hemisphere divided by alpha power measured from the left brain hemisphere. A ratio higher than 1 (1 infers that both sides of the brain are equal) correlates with depression.
Time Frame: Baseline, Post-TMS, 1-month and 6-month follow-up
Population: Subject 1: post-TMS HD-EEG data file is not retrievable. Subject 3 and 4: baseline and post-TMS data were too noisy for analysis in frequency domain, and therefore, were excluded from the following analysis.
  6-month follow-up: was not collected for this outcome measure due to COVID-19 pandemic
Measure: Mean (Standard Deviation); unit: frontal alpha power ratio R/L
Arm/Group | Low Frequency TMS Intervention
Number analyzed (Participants) | 10
frontal alpha power ratio R/L
  Baseline alpha power asymmetry | 1.29 (0.88)
  Post-TMS alpha power asymmetry: number analyzed (Participants) | 9
  Post-TMS alpha power asymmetry | 1.10 (0.21)
  1-Month Follow-up alpha power asymmetry: number analyzed (Participants) | 9
  1-Month Follow-up alpha power asymmetry | 1.35 (0.53)

5. Secondary Outcome: Changes in Depression Severity Related to the Study Interventions.
Description: Exploratory analyses will investigate changes in depression scores as a result of the study protocol and interventions. Quick Inventory of Depressive Symptomology (QIDS) is a self-assessment questionnaire used in this study to measure participants' depression symptoms. For Major Depressive Disorder scores of 0-5 indicate no depression, 6-10 indicates mild depression, 11-15 is moderate depression, 16-20 is severe depression, and 21-27 is very severe depression.
Time Frame: 1-week post-treatment, 1-month post-treatment, 3-month post-treatment, and 6-month post-treatment follow-up
Population: 3-month follow-up: subjects 1 & 2: data not available as this was not in the protocol at the time 6-month follow-up: subjects 3, 9, 13, 14: lost to follow-up, no data available for analysis
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Low Frequency TMS Intervention
Number analyzed (Participants) | 12
score on a scale
  Screening Visit | 16.9 [9 to 21]
  1-week post treatment | 8.2 [2 to 15]
  1-month post treatment | 8.7 [3 to 17]
  3-month post-treatment: number analyzed (Participants) | 10
  3-month post-treatment | 8.8 [3 to 19]
  6-month post-treatment: number analyzed (Participants) | 8
  6-month post-treatment | 9.6 [3 to 14]

ADVERSE EVENTS:
Time Frame: The adverse events are collected from each participant beginning at the screening visit up to the 6-month follow up visit. The results are expressed as the total number of adverse events recorded from all participants at the above specific study timeframe.
Arm/Group | Low Frequency TMS Intervention
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 12/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Frequency TMS Intervention (N=12)
Lower Back Pain (Musculoskeletal and connective tissue disorders) | 2
Mild Headache (General disorders) | 11
Eye Pain (General disorders) | 4
Fatigue (General disorders) | 3
Nausea (Gastrointestinal disorders) | 1
Bilateral Ear Discomfort (General disorders) | 1
Blurry Vision (General disorders) | 1
Lightheadedness (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-10-25): https://cdn.clinicaltrials.gov/large-docs/00/NCT03105700/Prot_SAP_000.pdf
  • Informed Consent Form (2020-09-24): https://cdn.clinicaltrials.gov/large-docs/00/NCT03105700/ICF_001.pdf